CLINICAL TRIAL: NCT01773902
Title: High Versus Standard Dose Protein for Very Preterm Infants
Brief Title: Protein for Premies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Axel Franz, PD Dr. med., University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PfP3.2
Record Dates: First submitted 2013-01-15; First posted 2013-01-23 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Extreme Prematurity
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High Dose Protein (Individualized) (Experimental): Protein supplementation according to breast milk content aiming for 4.5g/kg/d of enteral protein if <1500g b.w. or 4.0g/kg/d of enteral protein if >1500g b.w. until 1 week before discharge
  Interventions: Dietary Supplement: High Dose Protein (Individualized)
- High Dose Protein (Standardized) (Experimental): Protein supplementation independent of individual breast milk content using a new high-dose-protein breast milk fortifier until 1 week before discharge
  Interventions: Dietary Supplement: High Dose Protein (Standardized)
- Standard protein supplementation (Active Comparator): Protein supplementation independent of individual breast milk content using a standard dose of a standard breast milk fortifier until 1 week before discharge
  Interventions: Dietary Supplement: Standard Protein Supplementation

INTERVENTIONS:
Dietary Supplement: High Dose Protein (Individualized) — Protein supplementation according to breast milk content aiming for 4.5g/kg/d of enteral protein if <1500g b.w. or 4.0g/kg/d of enteral protein if >1500g b.w. until 1 week before discharge
  Arms: High Dose Protein (Individualized)
Dietary Supplement: High Dose Protein (Standardized) — Protein supplementation independent of individual breast milk content using a new high-dose-protein breast milk fortifier until 1 week before discharge
  Arms: High Dose Protein (Standardized)
Dietary Supplement: Standard Protein Supplementation — Protein supplementation independent of individual breast milk content using a standard-dose-protein breast milk fortifier until 1 week before discharge
  Arms: Standard protein supplementation

SUMMARY:
Although expressed breast milk is considered the optimal nutritional source for preterm infants, the macronutrient content is insufficient to enable optimal growth during neonatal intensive care. Optimal dose and optimal mode of administration (standardized or individualized) of enteral protein supplementation to very preterm infants have not been established.

This study aims to compare the effects on weight gain of different modes of enteral protein supplementation.

ELIGIBILITY:
Inclusion Criteria:

* very preterm infants <32 weeks gestation and <1500g birth weight
* > 100ml/kg/d of enteral feeding

Exclusion Criteria:

* missing informed consent
* decision not to feed breast milk
* congenital malformations
* age > 7 days at study entry

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Weight gain | From birth - to the end of study intervention (anticipated to be on average 1 week before discharge home at approx 37 weeks PMA)

SECONDARY OUTCOMES:
Head circumference growth | From birth - to the end of study intervention (anticipated to be on average 1 week before discharge home at approx 37 weeks PMA)

OTHER OUTCOMES:
Plasma amino acid profile | at 2 and 4 weeks after start of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Axel Franz, MD, Principal Investigator — Universität Tübingen
Locations (1):
- University Children's Hospital Tuebingen, Tübingen, Germany

REFERENCES:
- [Result] Maas C, Mathes M, Bleeker C, Vek J, Bernhard W, Wiechers C, Peter A, Poets CF, Franz AR. Effect of Increased Enteral Protein Intake on Growth in Human Milk-Fed Preterm Infants: A Randomized Clinical Trial. JAMA Pediatr. 2017 Jan 1;171(1):16-22. doi: 10.1001/jamapediatrics.2016.2681. PMID 27893064
- [Derived] Mathes M, Maas C, Bleeker C, Vek J, Bernhard W, Peter A, Poets CF, Franz AR. Effect of increased enteral protein intake on plasma and urinary urea concentrations in preterm infants born at < 32 weeks gestation and < 1500 g birth weight enrolled in a randomized controlled trial - a secondary analysis. BMC Pediatr. 2018 May 8;18(1):154. doi: 10.1186/s12887-018-1136-5. PMID 29739389
- [Derived] Maas C, Franz AR, Shunova A, Mathes M, Bleeker C, Poets CF, Schleicher E, Bernhard W. Choline and polyunsaturated fatty acids in preterm infants' maternal milk. Eur J Nutr. 2017 Jun;56(4):1733-1742. doi: 10.1007/s00394-016-1220-2. Epub 2016 May 10. PMID 27164830